CLINICAL TRIAL: NCT00000444
Title: Timing of Smoking Intervention in Alcohol Treatment
Brief Title: Timing of Smoking Intervention in Alcohol Treatment (Nicotine Patch)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAJOS11124; R01AA011124 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Alcoholism; Smoking
MeSH Terms: conditions — Alcoholism; Smoking | interventions — Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: nicotine replacement patch

SUMMARY:
This study will attempt to determine the best time to begin a smoking cessation program in individuals who undergo intensive treatment for alcohol dependence. The goal of this trial is to determine whether a smoking cessation program is more effective if it occurs at the same time as or after treatment for alcohol dependence. The study also will attempt to determine the effect of smoking cessation programs on the outcome of treatment for alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol use disorder and other drug dependence.
* Complete first week of alcohol treatment program.
* Current cigarette smoker (more than 5 cigarettes/day, smoking more than 1 year).

Exclusion Criteria:

* Lifetime diagnosis of an excluding psychiatric disorder: bipolar disorder, schizophrenia or other psychotic disorder, panic disorder with or without agoraphobia, obsessive-compulsive disorder, generalized anxiety disorder, eating disorder, post- traumatic stress disorder, antisocial personality disorder, or borderline personality disorder.
* Unable to participate in protocol due to functional deficits or severe depression.
* Suicidal or homicidal ideation.
* Current use of disulfiram (Antabuse) or naltrexone (Revia).
* Current use of pipes, cigars, or smokeless tobacco and unwillingness to stop.
* Lives more than 100 miles from alcohol treatment facility.
* No telephone.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1997-09; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- General Internal Medicine, VA Medical Center, Minneapolis, Minnesota, United States